CLINICAL TRIAL: NCT06212518
Title: Transdermal Optical Imaging (TOI) as a Non-invasive Measure to Detect Changes in Hydration Status in Healthy Adults and Athletes: Phase 3b Multi-center Trial for Model Development
Brief Title: Transdermal Optical Imaging (TOI) as a Non-invasive Measure to Detect Changes in Hydration Status in Healthy Adults and Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PEP-2306 3b
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Dehydration
Keywords: hydration; dehydration; euhydration; hypohydration; exercise; Transdermal Optical Imaging; TOI
MeSH Terms: conditions — Dehydration; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GENPOP passive dehydration (Experimental): In the 24 hours between the first and last face scan, reduce fluid intake by approximately 75% (equating to approximately 700 ml (women) and 800 ml (men)). Participants will be provided pre-filled water bottles and asked to only ingest fluid in bottle until second morning face scan.
  Interventions: Other: GENPOP fluid restriction
- GENPOP ad libitum fluid intake (Experimental): No fluid restriction
  Interventions: Other: GENPOP ad libitum fluid intake
- ATHLETE with fluid restriction (Experimental): For 24 hours prior to the study session, encouraged to drink sufficient fluid to maintain euhydration. Asked to refrain from alcohol 24 hours prior to session. Not permitted to drink during training session.
  Interventions: Other: ATHLETE restricted fluid intake
- ATHLETE ad libitum fluid intake (Experimental): For 24 hours prior to the study session, encouraged to drink sufficient fluid to maintain euhydration. Asked to refrain from alcohol 24 hours prior to session. Permitted to drink during training session.
  Interventions: Other: ATHLETE ad libitum fluid intake

INTERVENTIONS:
Other: GENPOP ad libitum fluid intake — Unrestricted fluid intake.
  Arms: GENPOP ad libitum fluid intake
Other: GENPOP fluid restriction — In the 24 hours between the first and last face scan, reduce fluid intake by approximately 75% (equating to approximately 700 ml (women) and 800 ml (men)).
  Arms: GENPOP passive dehydration
Other: ATHLETE ad libitum fluid intake — No restriction on fluid intake
  Arms: ATHLETE ad libitum fluid intake
Other: ATHLETE restricted fluid intake — Not permitted to drink during training session.
  Arms: ATHLETE with fluid restriction

SUMMARY:
The primary objective of this study is to analyze smart phone-based Transdermal Optical Imaging (TOI) features to develop a model that can discern hydration status, including: 1) at various timepoints throughout a 24-hour period in healthy adults from the general population (GENPOP), and 2) before and after a team coach-led training session in athletes competing in a sport (ATHLETE). TOI data will be collected alongside standard reference measures of hydration status.

In this study each subject will serve as their own control.

ELIGIBILITY:
Inclusion Criteria:

Both Study Arms (GENPOP and ATHLETE)

* Subject is male or female
* If female, subject is not pregnant
* Subject is willing to avoid alcohol consumption 24 hours prior to visit(s)
* Subject is willing to avoid wearing makeup to the study session or willing to remove it with facial wipes before the face scans
* Subject is willing to shave facial hair if predetermined during the informed consent session it will interfere with TOI measurement
* Able to speak, write, and read English
* Provision of written consent to participate

GENPOP Study

* Study subject is 18-65 years of age, inclusive
* Subject does not smoke (or has quit for at least 6 months)
* Subject is not taking medication that may interfere with the study
* Subject has no health conditions that would prevent completion of the trial as indicated on the general health questionnaire (GHQ)
* Subject is willing to fast overnight (~8-12 hours)
* Subject is willing to refrain from vigorous exercise for 48 hours
* Subject is willing to eat the exact same food the day prior to each visit to the testing site

ATHLETE Study

* Study subject is 14-45 years of age, inclusive
* Subject is participating in team sport training/competition
* Subject is participating in a coach-led practice

Exclusion Criteria:

Both Study Arms (GENPOP and ATHLETE)

* Subject has participated or currently enrolled in a clinical trial within the past 30 days
* Subject has participated in any PepsiCo trial within past 6 months
* Subject has a condition or is taking medication that the investigator believes would interfere with his/her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the person at undue risk
* Subject is allergic to alcohol or facial cleansing wipes
* Subject is employed by, or has a parent, guardian, or other immediate family member employed by a company that manufactures any products that compete with any Gatorade product. If subject is unsure if a company would be considered a competitor to Gatorade, they will be asked to please let the study investigator know the name of the other company and the nature of their relationship to that company before they sign the informed consent.

GENPOP Study

• Subject has a health condition or is taking medication that can be worsened by fluid restriction (participants who opt-in to fluid restriction study arm only)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Transdermal Optical Imaging (TOI) signals | Four time points for GENPOP over 24 hours (Day 1 ~8 a.m., ~11:30 a.m., ~3:30 p.m., Day 2 ~8.a.m.; for ATHLETES, on arrival before a single ~45 minute exercise training session and immediately following a 30 minute cool down period post-exercise
  Blood flow patterns of the face obtained from the video camera on a smart phone
Standard measurement of hydration status: Body mass change | Four time points for GENPOP over 24 hours (Day 1 ~8 a.m., ~11:30 a.m., ~3:30 p.m., Day 2 ~8.a.m.; for ATHLETES, upon arrival before a single ~45 minute exercise training session and again immediately after exercise
  Body mass scale (Tanita, WB-800 Plus) to the nearest 0.01 kilogram (kg)
Standard measurements of hydration status: Urine specific gravity | Four time points for GENPOP over 24 hours (Day 1 ~8 a.m., ~11:30 a.m., ~3:30 p.m., Day 2 ~8.a.m.; for ATHLETES, upon arrival before a single ~45 minute exercise training session and again immediately after exercise
  Digital pen refractometer (Atago, PEN-Urine SG)
Standard measurements of hydration status: Urine color | Four time points for GENPOP over 24 hours (Day 1 ~8 a.m., ~11:30 a.m., ~3:30 p.m., Day 2 ~8.a.m.; for ATHLETES, upon arrival before a single ~45 minute exercise training session and again immediately after exercise
  Color range scale rated from dilute to concentrated. 1=clear through yellows and oranges with most orange =7
Standard measurements of hydration status: Thirst | Four time points for GENPOP over 24 hours (Day 1 ~8 a.m., ~11:30 a.m., ~3:30 p.m., Day 2 ~8.a.m.; for ATHLETES, on arrival before a single ~45 minute exercise training session and immediately following a 30 minute cool down period post-exercise
  Categorical scale from 1=Not thirsty at all, to 7=very, very thirsty

SECONDARY OUTCOMES:
Subject demographics - Age | At screening
  in years
Subject demographics - Sex | At screening
  male or female
Subject demographics - Ethnicity | At screening
  Hispanic or Latino, or not Hispanic or Latino
Subject demographics - Race | At screening
  American Indian, Alaska native, Asian, Black or African American, Native Hawaiian or Pacific Islander, White
Fitzpatrick classification of skin color | At screening
  Skin type from 1=White skin, always burns, never tans to 6 = Black skin, heavily pigmented, never burns, tans very easily
Mood scale | Four time points for GENPOP over 24 hours (Day 1 ~8 a.m., ~11:30 a.m., ~3:30 p.m., Day 2 ~8.a.m.; for ATHLETES, on arrival before a single ~45 minute exercise training session and immediately following a 30 minute cool down period post-exercise
  Rated from 1=Calm to 9=Irritated
Dietary and fluid intake | For GENPOP from 24 hours prior to Day 1 visit (~8 a.m.) through end of testing period (Day 2 ~8 a.m.). For ATHLETES from 24 hours to prior to start of single ~45 minute exercise session (if fluid restricted) or to end of exercise (if ad lib fluid intake)
  Food and fluid intake recorded on a paper log

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Baker, PhD, Study Director — PepsiCo, Inc. Sports Science; Matt Hinkley, PhD, Principal Investigator — Pepsico, Inc. Sports Science
Locations (4):
- United States (4):
  - Pepsico R&D Life Sciences, Bradenton, Florida
  - PepsiCo R&D Gatorade Sports Science Institute, Chicago, Illinois
  - PepsiCo R&D, Gatorade Sports Science Institute, Valhalla, New York
  - PepsiCo R&D, Gatorade Sports Science Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No